CLINICAL TRIAL: NCT06384404
Title: Functional Outcomes in Patients Who Undergo Upfront Surgical Resection for High-Grade Osteosarcoma of the Extremity: A Pilot Study
Brief Title: Upfront Surgical Resection for Osteosarcoma
Acronym: UFSR for OS
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-14741
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteosarcoma: Patients with newly diagnosed osteosarcoma
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — PROMIS questionnaire

SUMMARY:
The goal of this pilot study is to learn about patients with newly diagnosed osteosarcoma of an extremity, and whether surgically removing the tumor prior to the administration of any chemotherapy will improve functional outcomes. In order to learn about the patient's experience, the study team will administer questionnaires to the patient and surgeon at various timepoints to assess recovery and the function of the extremity.

DETAILED DESCRIPTION:
This prospective, non-randomized pilot study will assess patient-reported functional outcomes of upfront surgical resection in patients with newly diagnosed, biopsy-proven, localized osteosarcoma of the extremity or the pelvis. Following biopsy, all patients will undergo wide excision of the tumor followed by systemic multi-agent cytotoxic chemotherapy consisting of a regimen at least equivalent to the standard of care of high dose Methotrexate, Doxorubicin, and Cisplatin (MAP). Patients and/or their parent/guardian will be administered PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaires, while surgeons will be administered the Musculoskeletal Tumor Society (MSTS) questionnaire at various timepoints through the first year post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed, previously untreated, localized, high-grade osteosarcoma of an extremity (verified by histopathology) with plans to undergo upfront surgical resection of the tumor followed by systemic chemotherapy.
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2 (Karnofsky will be used for patients >16 years of age and Lansky score for patients <= 16 years of age)

Exclusion Criteria:

* Patients with metastatic disease at diagnosis
* Initiation of systemic therapy prior to enrollment
* Prior history of cancer
* Prior radiation therapy
* Active life-threatening infection
* Pregnancy (negative pregnancy test result must be obtained for female patients of childbearing potential)

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with newly diagnosed osteosarcoma with plans to undergo an upfront surgical resection of their tumor.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (HRQoL) score from Historical Controls | approximately 1 year
  Modified age-based PROMIS measures will be used to assess HRQoL changes (PROMIS 25 Parent Proxy will be used for ages 5-7; PROMIS 25 for 8-17; PROMIS 29+2 for 18+)
  PROMIS 25 (and PROMIS 25 Parent Proxy) contain six, 4-item short forms for domains: physical function mobility, anxiety, depressive symptoms, fatigue, peer relationships, pain interference; along with a pain intensity item. Scores for each domain range from 1-5 (pain intensity 0-10). Responses to individual items are coded to values and summed to generate a total raw score. Total raw scores are converted/rescaled into a standardized T-score for each participant with a mean of 50 and a standard deviation (SD) of 10. Higher PROMIS T-scores represent more of the concept being measured
  PROMIS 29+2 is similar to PROMIS 25 with the exception of a social roles/activities domain in place of peer relationships, and also includes sleep disturbance and cognitive function domains. Scores are determined as described for PROMIS 25

SECONDARY OUTCOMES:
Event Free Survival | Up to 2 years
  The number of participants with event-free survival (EFS) will be determined. Event-free survival will be defined as the time from diagnosis until disease progression, recurrence at any site, secondary malignancy, death, or last follow-up, whichever is observed first

CONTACTS AND LOCATIONS:
Overall Officials: Alice Lee, M.D., Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Imran H, Enders F, Krailo M, Sim F, Okuno S, Hawkins D, Neglia J, Randall RL, Womer R, Mascarenhas L, Arndt CA. Effect of time to resumption of chemotherapy after definitive surgery on prognosis for non-metastatic osteosarcoma. J Bone Joint Surg Am. 2009 Mar 1;91(3):604-12. doi: 10.2106/JBJS.H.00449. PMID 19255220
- [Background] Link MP, Goorin AM, Miser AW, Green AA, Pratt CB, Belasco JB, Pritchard J, Malpas JS, Baker AR, Kirkpatrick JA, et al. The effect of adjuvant chemotherapy on relapse-free survival in patients with osteosarcoma of the extremity. N Engl J Med. 1986 Jun 19;314(25):1600-6. doi: 10.1056/NEJM198606193142502. PMID 3520317
- [Background] Xu J, Xie L, Guo W. Neoadjuvant Chemotherapy Followed by Delayed Surgery: Is it Necessary for All Patients With Nonmetastatic High-Grade Pelvic Osteosarcoma? Clin Orthop Relat Res. 2018 Nov;476(11):2177-2186. doi: 10.1097/CORR.0000000000000387. PMID 29912746
- [Background] Reed DR, Metts J, Pressley M, Fridley BL, Hayashi M, Isakoff MS, Loeb DM, Makanji R, Roberts RD, Trucco M, Wagner LM, Alexandrow MG, Gatenby RA, Brown JS. An evolutionary framework for treating pediatric sarcomas. Cancer. 2020 Jun 1;126(11):2577-2587. doi: 10.1002/cncr.32777. Epub 2020 Mar 16. PMID 32176331
- [Background] Hinds PS, Gattuso JS, Billups CA, West NK, Wu J, Rivera C, Quintana J, Villarroel M, Daw NC. Aggressive treatment of non-metastatic osteosarcoma improves health-related quality of life in children and adolescents. Eur J Cancer. 2009 Jul;45(11):2007-14. doi: 10.1016/j.ejca.2009.04.020. Epub 2009 May 18. PMID 19450974
- [Background] Bell RS, Roth YF, Gebhardt MC, Bell DF, Rosenberg AE, Mankin HJ, Suit HD. Timing of chemotherapy and surgery in a murine osteosarcoma model. Cancer Res. 1988 Oct 1;48(19):5533-8. PMID 3166399